CLINICAL TRIAL: NCT03168516
Title: Effects of Closed-loop Automatic Control of the Inspiratory Fraction of Oxygen (FiO2-C) on Outcome of Extremely Preterm Infants - a Randomized Controlled Parallel Group Multicenter Trial for Safety and Efficacy
Brief Title: Effects of Closed-loop Automatic Control of FiO2 in Extremely Preterm Infants
Acronym: FiO2-C
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FiO2-C; 2018-000453-41 (EudraCT Number); BMBF-Fz01KG1602 (Other Grant/Funding Number: BMBF)
Record Dates: First submitted 2017-05-18; First posted 2017-05-30 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-07

CONDITIONS: Infant,Premature
Keywords: Oxygen; closed-loop automatic control; Oxygen saturation; preterm infants
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental intervention (Experimental): closed-loop automatic control of the inspiratory fraction of oxygen (FiO2-C)
  Interventions: Device: closed-loop automatic control of the inspiratory fraction of oxygen (FiO2-C)
- Control intervention (No Intervention): Standard care, i.e. manual adjustments of the FiO2 only

INTERVENTIONS:
Device: closed-loop automatic control of the inspiratory fraction of oxygen (FiO2-C) — Application of FiO2-C (provided by standard infant ventilators) in addition to manual adjustments of the inspired oxygen fraction (FiO2) during mechanical ventilation and continuous positive airway pressure (CPAP) in ELGANs at least up to 32weeks PMA according to a standardized protocol
  Arms: Experimental intervention

SUMMARY:
Extremely low gestational age neonates (ELGANs), i.e. those born at <28 weeks, frequently experience intermittent hypoxemic/hyperoxemic episodes. Observational data indicate that severe and prolonged hypoxemic episodes are associated with retinopathy of prematurity (ROP), impaired long-term development and death. Closed-loop automated control of the inspiratory fraction of oxygen (FiO2-C) reduces time outside the oxygen target range, decreases number and duration of hypo- and hyperoxemic episodes, and reduces caregivers' workload. The proposed observer-blinded randomized controlled trial was designed and will be powered to compare the effect of FiO2-C in addition to manual adjustments, in comparison with manual adjustments of FiO2 only, on death and severe complications of prematurity thought to be related to hypoxia/hyperoxia and neurodevelopmental impairment in ELGANs. The results of this trial may help to improve the quality of life of ELGANs and reduce the burden of significant morbidity as well as costs for health care and society

DETAILED DESCRIPTION:
Approximately 0.5% of all neonates (i.e., about 25,000 infants per year in Europe) are extremely low gestational age neonates (ELGANs), i.e. have a gestational age (GA) of <28 completed weeks at birth. ELGANs have higher incidences of mortality, retinopathy of prematurity (ROP), chronic lung disease and other risks of prematurity as well as severe neurodevelopmental impairment.

The vast majority of ELGANs require supplemental oxygen in addition to mechanical respiratory support (including CPAP). Irrespective of the SpO2 target, the vast majority of ELGANs suffers from recurrent intermittent hypoxemic and (as a consequence of inappropriate adjustments of FiO2) hyperoxemic episodes. Recurrent intermittent hypoxic episodes - i.e. wide fluctuations in oxygen levels - are associated with an increased risk of ROP and there are data that suggest that late deaths and neurodevelopmental impairment are also linked to them.

Continuous positive airway pressure (CPAP) has been shown to reduce extubation failure in preterm infants, which may in part be due to a reduced frequency and severity of apnea of prematurity and stabilized functional residual capacity during apnea. Keeping oxygen levels (i.e., SpO2) stable despite irregular breathing patterns in ELGANs, requires frequent adjustments of the FiO2 which is both challenging, time consuming, and often impossible due to limited personnel resources.

FiO2-Controllers have been developed by several manufacturers of infant ventilators. They reduce the burden of hyper-/hypoxemia in infants while being safe and accurate in very short-term studies. The effects of FiO2-C on clinically relevant outcome measures and the safety of long-term continuous application, however, have yet to be elucidated. Hence there is now a window of opportunity to assess this new technology for benefits and harms, before it is implemented into neonatal care without appropriate evaluation of its safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants with a gestational age (GA) at birth of 23+0/7 - 27+6/7 weeks

Exclusion Criteria:

* Decision for palliative care
* congenital anomalies
* postnatal age > 48h
* missing parental consent
* lack of device enabling closed-loop automatic control of FiO2

Max Age: 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1065 (Actual)
Dates: Start 2018-07-27 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Primary outcome I: composite outcome of death, severe retinopathy of prematurity (ROP), chronic lung disease of prematurity (BPD), necrotizing enterocolitis (NEC) | until/at post-menstrual age (PMA) 36 weeks (death, BPD and NEC) and at latest at PMA 44 weeks for severity of ROP
  The primary outcome I is a composite of any of the following:
  * Death
  * Severe retinopathy of prematurity (severe ROP, as defined in 7.3.1)
  * Chronic lung disease of prematurity (BPD, according to the physiological definition, which is described in detail in the study protocol)
  * Necrotizing enterocolitis (NEC, as defined in the study protocol) until discharge from hospital
  The primary endpoint I will be analysed between the two intervention groups using a stratified chi2-test and Cochrane Mantel-Haenszel statistics will be presented (risk ratios and 95%-confidence intervals). The factors considered for randomization (center, sex and gestational age at birth (<26 weeks and ≥26 weeks) will also be used for analysis.
Primary outcome II: composite of death or neurodevelopmental impairment (NDI) | at 24 months of age corrected for prematurity
  The primary outcome II is a composite of any of the following:
  • death or neurodevelopmental impairment (defined as at least one of the following components: motor disability (GMFCS 2-5), language or cognitive delay (language composite score < 85 or cognitive composite score < 85 on Bayley Scales of Infant Development, 3rd edition) or severe visual or hearing impairment (need for a hearing aid or cochlear implant)). In case of missing Bayley III test results, Bayley II results, other developmental test results or PARCA-R parent questionnaire results may substitute for the Bayley III test results in a hierarchical manner described in the study protocol.
  The primary outcome II will be analysed between the two intervention groups using chi2-test and Cochrane Mantel-Haenszel statistics will be presented (risk ratios and 95%-confidence intervals). The factors considered for randomization (center, sex and gestational age at birth (<26 weeks and ≥26 weeks) will also be used for analysis.

SECONDARY OUTCOMES:
Death | 24 months of age corrected for prematurity
  Death rates will be compared between the two treatment groups and analyzed by Cochrane-Mantel-Haenszel- X²-Test.
ROP Severity Score | at latest at PMA 44 weeks
  The most severe grade of ROP according to 25 categories currently developed by the working group of the international neonatal consortium (may have to be adapted as the consensus process proceeds), documented in either eye (for at least 2 consecutive examinations) will be analysed using Wilcoxon-Mann-Whitney test.
Severe ROP | at latest at PMA 44 weeks
  defined as: ROP stage 0, 1 or 2 (in Zone 2 or 3) = no/non-severe ROP versus 3, 4 or 5, or AP-ROP, or any ROP in Zone 1, or any treatment for ROP = severe ROP.
  Rates of severe ROP will be compared between the two treatment groups and analyzed by Cochrane-Mantel-Haenszel- X²-Test.
bronchopulmonary Dysplasia (BPD) | until 36 weeks PMA
  As part of routine care, the presence of BPD will be determined at 36 weeks postmenstrual age (PMA) according to the physiological definition of Walsh et al. [Walsh, J Perinatol 2003].
  BPD rates will be compared between the two treatment groups and analyzed by Cochrane-Mantel-Haenszel- X²-Test.
Necrotizing enterocolitis (NEC) | until 36 weeks PMA
  NEC (modified Bell stage ≥ IIA according to [Bell, Ann Surg 1978]) or intestinal perforation will be diagnosed at surgery, at autopsy, or by either the finding of pneumatosis intestinalis, hepatobiliary gas, or free intraperitoneal air on abdominal x-ray, or by demonstration of gas (bubbles) in the portal vein on abdominal ultrasound or abdominal x-ray.
  NEC rates will be compared between the two treatment groups and analyzed by Cochrane-Mantel-Haenszel- X²-Test.
Neurodevelopmental impairment (NDI) | at 24 months of age corrected for prematurity
  NDI is defined as at least one of the following components: motor disability (modified GMFCS 2-5), language or cognitive delay (language composite score < 85 or cognitive composite score < 85 on Bayley Scales of Infant Development, 3rd edition) or severe visual or hearing impairment (need for a hearing aid or cochlear implant).
  In case of missing Bayley III test results, Bayley II results, other developmental test results or PARCA-R parent questionnaire results may substitute for the Bayley III test results in a hierarchical manner described in the study protocol.
  NDI rates will be compared between the two treatment groups and analyzed by Cochrane-Mantel-Haenszel- X²-Test.
Bayley III. Language composite score - dichotomized | at 24 months of age corrected for prematurity
  The results of the language composite score of the Bayley Scales of Infant Development, 3rd edition, will be dichotomized by <85 (abnormal) versus >=85 (normal) and compared between the two treatment groups by Cochrane-Mantel-Haenszel- X²-Test.
Bayley III: Language composite score - numerical | at 24 months corrected age
  The raw numerical data of the language-composite-score will be analysed using Wilcoxon-Mann-Whitney test. The use of this test accounts for the fact that data will be cut due to lack sensitivity below 50 points.
Bayley III: Cognitive composite score - dichotomized | at 24 months of age corrected for prematurity
  The results of the cognitive composite score of the Bayley Scales of Infant Development, 3rd edition, will be dichotomized by <85 (abnormal) versus >=85 (normal) and compared between the two treatment groups by Cochrane-Mantel-Haenszel- X²-Test.
Bayley III: Cognitive composite score - numerical | at 24 months of age corrected for prematurity
  The numerical data of the cognitive-composite-score will be analysed using Wilcoxon-Mann-Whitney test. The use of this test accounts for the fact that data will be cut due to lack sensitivity below 50 points.
Cerebral palsy | at 24 months of age corrected for prematurity
  Cerebral palsy will be diagnosed if the child has a non-progressive motor impairment characterized by abnormal muscle tone and impaired range or control of movements, according to the criteria defined by the European network 'Surveillance of CP in Europe'.
  Rates of cerebral palsy will be compared between the two treatment groups and analyzed by Cochrane-Mantel-Haenszel- X²-Test.
Motor disability | at 24 months of age corrected for prematurity
  Motor disability is defined as a modified GMFCS 2-5 versus a modified GMFCS 0-1, which is regarded as being normal. Rates of motor disability will be compared between the two treatment groups and analyzed by Cochrane-Mantel-Haenszel- X²-Test.
Score data of modified Gross Motor Function Classification Scale (GMFCS) | at 24 months of age corrected for prematurity
  GMFCS-Score for quantification of the effects of cerebral palsy and other motor impairments (adapted from Palisano et al. [Palisano Med Child Neurol 1997]) using the FiO2-C-GMFCS-score sheet (separate document not part of this protocol) will be analysed. GMFCS-score consists of six categories. Analysis will be done by using Wilcoxon-Mann-Whitney test.
Bayley III: Motor composite score - numerical | at 24 months of age corrected for prematurity
  The numerical data of the motor-composite-score will be analysed using Wilcoxon-Mann-Whitney test. The use of this test accounts for the fact that data will be cut due to lack of sensitivity below 50 points.
Severe visual impairment | at 24 months of age corrected for prematurity
  Severe visual impairment is defined as an ophthalmological assesment indicating "severe visual impairment", e.g. the best corrected vision in the better eye yields a visual acuity less than 6/60 m (20/200 ft).
  Rates will be compared between the two treatment groups and analyzed by Cochrane-Mantel-Haenszel- X²-Test.
Severe hearing impairment | at 24 months of age corrected for prematurity
  Severe hearing impairment is defined as need for a hearing aid or cochlear implant. Rates will be compared between the two treatment groups and analyzed by Cochrane-Mantel-Haenszel- X²-Test.

CONTACTS AND LOCATIONS:
Overall Officials: Axel Franz, Prof. Dr., Study Director — University Children's Hospital Tuebingen
Locations (32):
- Northwest Women's and Children's Hospital, Xi'an, China
- Germany (27):
  - Klinikum St. Marien - Klinik für Kinder und Jugendliche, Amberg
  - Josefinum - Klinik für Kinder und Jugendliche, Augsburg
  - Diakonie Krankenhaus der Kreuznacher Diakonie, Bad Kreuznach
  - Klinikum Links der Weser, Bremen
  - Universitätsklinikum Dresden, Dresden
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - HELIOS Klinikum Erfurt, Erfurt
  - Klinikum Esslingen GmbH - Klinik für Kinder und Jugendliche, Esslingen am Neckar
  - Zentrum für Kinder- und Jugendmedizin, Freiburg im Breisgau
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - Städtisches Klinikum Karlsruhe, Karlsruhe
  - University Hospital Leipzig, Leipzig
  - Städtisches Klinikum - Klinik für Neonatologie, München
  - München Klinik Harlaching, München
  - Universitätsklinikum München, München - Großhadern
  - Klinik für Kinder- und Jugendmedizin, Münster
  - Klinik Hallerwiese - Cnopf'sche Kinderklinik, Nuremberg
  - Krankenhaus Barmherzige Brüder, Regensburg
  - Klinikum am Steinenberg, Reutlingen
  - Leopoldina Krankenhaus der Stadt Schweinfurt GmbH, Schweinfurt
  - Diakonissen-Stiftungs-Krankenhaus Speyer, Speyer
  - Klinikum Stuttgart, Olgahospital, Stuttgart
  - University Hospital Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm
  - Schwarzwald-Baar-Klinik, Villingen-Schwenningen
  - Rems-Murr-Kliniken gGmbH, Winnenden
- Netherlands (3):
  - Kindergeneeskunde Maastricht Universitair Medisch Centrum, Maastricht
  - Máxima Medical Center, Veldhoven
  - Isala Kliniek Zwolle - Location Sophia, Zwolle
- The James Cook University Hospital, Middlesbrough, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Maiwald CA, Niemarkt HJ, Poets CF, Urschitz MS, Konig J, Hummler H, Bassler D, Engel C, Franz AR; FiO2-C Study Group. Effects of closed-loop automatic control of the inspiratory fraction of oxygen (FiO2-C) on outcome of extremely preterm infants - study protocol of a randomized controlled parallel group multicenter trial for safety and efficacy. BMC Pediatr. 2019 Oct 21;19(1):363. doi: 10.1186/s12887-019-1735-9. PMID 31630690
- [Derived] Konig J, Stauch A, Engel C, Urschitz MS, Franz AR; FiO2-C study group. Statistical analysis plan for the FiO2-C trial: effects of closed-loop automatic control of the inspiratory fraction of oxygen (FiO2-C) on outcomes of extremely preterm infants-a randomized-controlled parallel group multicentre trial for safety and efficacy. Trials. 2024 Nov 12;25(1):756. doi: 10.1186/s13063-024-08615-7. PMID 39533330
- See also: study homepage — http://www.fioc-study.eu/